CLINICAL TRIAL: NCT06981221
Title: Predictors of Pleth Variability Index During Laparoscopically Assisted Vaginal Hysterectomy
Brief Title: PVI Predictors in Laparoscopic Hysterectomy
Status: Completed | Type: Observational
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor, Wonkwang University Hospital
Other Study IDs: Wonkwang UH19
Record Dates: First submitted 2025-05-07; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Hysterectomy; PVI; Fluid Responsiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Masimo Radical-7 Pulse Oximeter — "PVI is continuously monitored using the Masimo Radical-7 pulse oximetry device to evaluate respiratory variation in the plethysmographic waveform amplitude during laparoscopic-assisted vaginal hysterectomy (LAVH). No fluid intervention is applied; device use is for observational measurement of fluid responsiveness."
  Other Names: PVI (Pleth Variability Index)

SUMMARY:
This observational study investigates the predictors of Pleth Variability Index (PVI) changes in euvolemic patients undergoing laparoscopic-assisted vaginal hysterectomy (LAVH). The primary objective is to quantify changes in PVI (ΔPVI) across six intraoperative time points associated with positional shifts. Secondary objectives include identifying key predictors of significant PVI change (ΔPVI ≥ 5%), such as passive leg raising, Trendelenburg position, body mass index (BMI), and intraabdominal pressure. Additional variables including perfusion index, mean arterial pressure, bispectral index, skin temperature, age, and anesthetic agent will be evaluated as potential modulators. Findings aim to support individualized fluid management strategies in LAVH.

DETAILED DESCRIPTION:
This prospective, single-center observational cohort study evaluates dynamic intraoperative changes in the Pleth Variability Index (PVI) in 50 adult female patients undergoing elective laparoscopically assisted vaginal hysterectomy (LAVH) at Wonkwang University Hospital.

After establishing euvolemia with a 500 mL Volulyte preload (Fresenius Kabi GmbH) over 30-50 minutes, no further intraoperative fluid boluses are given. Anesthesia is induced with propofol (2 mg/kg), fentanyl (1-2 μg/kg), and rocuronium (0.6 mg/kg), and maintained with sevoflurane or desflurane titrated to a bispectral index (BIS) of 40-60. Pneumoperitoneum is set at 12-15 mmHg, and positional maneuvers include 30° passive leg raising, 15° Trendelenburg, and 15° reverse Trendelenburg.

Monitoring devices and data acquisition:

* **Masimo Radical-7** pulse oximeter (PVI, perfusion index [PI])
* **Invasive arterial line** (mean arterial pressure [MAP])
* **BIS sensor** (BIS)
* **Skin temperature probe** (forearm, °C) calibrated pre-case

Measurements are recorded at six standardized time points (baseline; post-induction; post-passive leg raising; post-pneumoperitoneum; post-Trendelenburg; post-reverse Trendelenburg). Continuous waveforms are averaged over 30 s epochs.

Primary endpoint is the absolute change in PVI (ΔPVI) relative to baseline. Secondary analyses include:

* Multivariable logistic regression for predictors of ΔPVI ≥ 5%
* Multivariable linear regression for continuous ΔPVI prediction
* Correlation analyses of ΔPVI with intraabdominal pressure (mmHg) and body mass index (kg/m²)
* Sensitivity analysis of PI reliability (intraclass correlation coefficient) across skin temperature thresholds
* Descriptive statistics for frequency of vasopressor (ephedrine) use

All analyses are performed using SPSS v29.0 with p < 0.05 considered statistically significant (Bonferroni correction applied for repeated measures).

ELIGIBILITY:
Inclusion Criteria:

* adult females aged 19-70 years (American Society of Anesthesiologists physical status I-III) scheduled for elective LAVH.

Exclusion Criteria:

* emergency surgery, severe cardiac or pulmonary disease, renal failure, pregnancy, or conditions contraindicating fluid administration. Participants were consecutively recruited during preoperative consultations.

Ages: 19 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult female patients aged 19 to 70 years with ASA physical status I-III who are scheduled to undergo elective laparoscopic-assisted vaginal hysterectomy (LAVH) at Wonkwang University Hospital. All participants are screened during routine preoperative consultations and provide written informed consent prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
ΔPVI (Change in Pleth Variability Index) | Intraoperative period (~60-90 minutes)
  Absolute change in PVI (%) at each of six intraoperative time points relative to baseline.

SECONDARY OUTCOMES:
Proportion of patients with significant ΔPVI ≥ 5% | At any of the six predefined intraoperative time points: • Post-induction • Post-passive leg raising • Post-pneumoperitoneum • Post-Trendelenburg • Post-reverse Trendelenburg • End of surgery (within 60-90 minutes after induction of anesthesia)
  Percentage of participants exhibiting a ΔPVI ≥ 5% at any intraoperative time point.
Effect of intraabdominal pressure on ΔPVI | At post-pneumoperitoneum and post-Trendelenburg time points (20-45 minutes after anesthesia induction)
  Correlation coefficient (r) between intraabdominal pressure (mmHg) and magnitude of ΔPVI.with magnitude of ΔPVI during pneumoperitoneum and Trendelenburg position. Multivariable linear regression is used.
Effect of body mass index on ΔPVI | ΔPVI measured at post-pneumoperitoneum and post-Trendelenburg time points (20-45 minutes after anesthesia induction)
  Correlation coefficient (r) between BMI (kg/m²) and magnitude of ΔPVI.measurements during LAVH. Data analyzed using subgroup comparison between stable and decreased skin temperature conditions.
Change in mean arterial pressure (MAP) | MAP measured at six predefined intraoperative time points: • Baseline • Post-induction • Post-passive leg raising • Post-pneumoperitoneum • Post-Trendelenburg • Post-reverse Trendelenburg (Total duration: ~90 minutes after anesthesia induction)
  Absolute change in MAP (mmHg) at the six predefined time points.
Change in perfusion index (PI) | MAP measured at six predefined intraoperative time points: • Baseline • Post-induction • Post-passive leg raising • Post-pneumoperitoneum • Post-Trendelenburg • Post-reverse Trendelenburg (Total duration: ~90 minutes after anesthesia induction)
  Absolute change in PI (unitless) at the six predefined time points.
Change in bispectral index (BIS) | MAP measured at six predefined intraoperative time points: • Baseline • Post-induction • Post-passive leg raising • Post-pneumoperitoneum • Post-Trendelenburg • Post-reverse Trendelenburg (Total duration: ~90 minutes after anesthesia induction)
  Absolute change in BIS (unitless) at the six predefined time points.
Influence of skin temperature on PI reliability | MAP measured at six predefined intraoperative time points: • Baseline • Post-induction • Post-passive leg raising • Post-pneumoperitoneum • Post-Trendelenburg • Post-reverse Trendelenburg (Total duration: ~90 minutes after anesthesia induction)
  Difference in intraclass correlation coefficient of PI measurements between stable (≤ ± 1 °C) and decreased (> 1 °C drop) skin temperature conditions.
Frequency of vasopressor use | MAP measured at six predefined intraoperative time points: • Baseline • Post-induction • Post-passive leg raising • Post-pneumoperitoneum • Post-Trendelenburg • Post-reverse Trendelenburg (Total duration: ~90 minutes after anesthesia induction)
  Number and percentage of patients requiring ephedrine bolus due to MAP < 70 mmHg during the observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Lee, M.D.,Ph.D, Study Director — Wonkwang University Hospital
Locations (1):
- Wonkwang University School of Medicine Hospital, Iksan, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided